CLINICAL TRIAL: NCT03625661
Title: Impact and Evaluation of the Management of Iron Deficiency With or Without Anemia in Patients With Cancer
Acronym: CAMARA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ICO-A-2013-07
Record Dates: First submitted 2018-07-04; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-07

CONDITIONS: Iron Deficiency Anemia
Keywords: Treatment Related Cancer,iron deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric carboxymaltose

STUDY DESIGN:
Intervention Model Description: cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm with Ferinject (Experimental): Ferinject will be administered once at inclusion
  Interventions: Drug: Ferinject

INTERVENTIONS:
Drug: Ferinject — Ferinject 50mg/ml, one injection
  Other Names: carboxymaltose ferrique

SUMMARY:
In oncology, anemia is a frequent symptom, leading to complication of patient management for, more or less, a long term but often poorly evaluated by medical teams.

In oncology, anemia is induced by multiple causes. Iron deficiency appears to be a leading cause of anemia, especially in people with solid cancer. Iron deficiency is characterized by a low level of iron . Iron is a trace element required for life. It is a major component of hemoglobin allowing the transport of oxygen in red blood cells. There are in fact 2 types of iron deficiency: an absolute iron deficiency with a deficiency of true iron and a functional iron deficiency. Since end of January 2014, intravenous iron-based injections have been reclassified for cancer patients at ICO Paul Papin. The monitoring of iron deficiency with or without anemia is currently done in our institute, the ICO-Paul Papin. There is a procedure for the management of anemia with or without iron deficiency but there is still no traceability of treatments performed, their compliance or even their impact on the rate hemoglobin and the quality of life of patients during their treatment. This observatory also makes it possible to evaluate the impact of this treatment on the quality of life of the patients and thus allows them a personalized care of the tiredness during their treatment

DETAILED DESCRIPTION:
The study is for patients with iron deficiency and / or anemia during treatment for cancer These patients will receive ferinject. Patients will perform functional assessments and complete quality of life questionnaires, when the ferinject will be injected, then at 1 month and 6 months.

Patients will be followed for 6 months in the study

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient with cancer regardless of the location
* Patient with specific treatment (chemotherapy +/- targeted therapy and / or radiotherapy, hormone therapy or surgery)
* Patient with Functional Iron Deficiency or absolute with or without anemia
* Having given written informed consent prior to any procedure related to the study.

Exclusion Criteria:

* Patient in a palliative situation not receiving specific treatment for their cancer
* Patient is willing and able to comply with the protocol for the duration of the study including all scheduled treatment, visits and examinations
* Patient with myeloproliferative disease
* Contraindication to treatments for iron deficiency and / or anemia
* Pregnant woman, parturient or nursing mothers
* Patient has no valid health insurance
* Disorder precluding understanding of trial information or informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2014-02-02 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-06-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the quality of life of patients with iron deficiency with or without anemia during treatment for their cancer | 42 months
  Obtained with the quality of life with the FACT-An questionnaire.

SECONDARY OUTCOMES:
Estimation of the proportion of absolute iron deficiency | 42 months
  Absolute iron deficiency is defined by a ferritin level <300 μg / L and a transferrin saturation coefficient <20%.
Estimation of the proportion of functional iron deficiency | 42 months
  Functional iron deficiency is defined by a ferritin level <800 μg / L and a Transferrin Saturation Coefficient <20%.
Estimation of the proportion of iron deficiency as a whole | 42 months
  Addition of proportion of iron deficiency
Estimation proportion of symptomatic anemia | 42 months
  Symptomatic anemia is defined as hemoglobin <12 g / dL associated with pallor and anoxic functional symptoms
Estimation of the proportion of asymptomatic anemia | 42 months
  Asymptomatic anemia is defined as hemoglobin <12 g / dL without clinical signs.
Estimation of the proportion of anemia as a whole | 42 months
  Addition of proportion of asymptomatic anemia and symptomatic anemia
Estimation of the proportion of undernourished patients | 42 months
  The diagnosis of malnutrition will be done by calculating BMI (<18.5 si - 70 years old and <21 from 70 years old)
Estimation of the evolution of the functional capacities of the patient | 42 months
  Estimated by functional questionnaire (Berg Balanced Scale test)
Estimation of the evolution of the functional capacities of the patient | 42 months
  Estimated by functional questionnaire (the Tinetti test)
Estimation of the evolution of the functional capacities of the patient | 42 months
  Estimated by functional questionnaire (the Timed Up and Go test)
Estimation of the evolution of the functional capacities of the patient | 42 months
  Estimated by functional questionnaire (the 6-minute walk test)
Estimation of the evolution of the functional capacities of the patient | 42 months
  Estimated by functional questionnaire (the 1-minute sit-stand test)
Estimation of the evolution of the functional capacities of the patient | 42 months
  Estimated by functional questionnaire (the climb and descent test of a staircase for 1 minute)

CONTACTS AND LOCATIONS:
Overall Officials: DELPHINE CORNUAULT-FOUBERT, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (1):
- Institut de Cancérologie de l'Ouest, Angers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gluszak C, de Vries-Brilland M, Seegers V, Baroin C, Kieffer H, Delva R, Cornuault-Foubert D. Impact of Iron-Deficiency Management on Quality of Life in Patients with Cancer: A Prospective Cohort Study (CAMARA Study). Oncologist. 2022 Apr 5;27(4):328-333. doi: 10.1093/oncolo/oyac005. PMID 35380718